CLINICAL TRIAL: NCT01045486
Title: A Double Blind, Randomized, Placebo-Controlled, Crossover Study to Compare the Effectiveness of Probiotics on Atopic Dermatitis With Cow Milk Allergy in Korean Infants
Brief Title: the Effectiveness of Probiotics on Atopic Dermatitis With Cow Milk Allergy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: failed to enroll patients
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Pediatric Allergy & Respiratory Center, Department of Pediatrics, Soonchunhyang University Hospital, Pediatric Allergy & Respiratory Center, Soonchunhyang University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: schprobiotics
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Food allergy; Probiotics
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Group A received active medication (ATP mixed probiotics) for 6 weeks followed by a crossover to 6 weeks of placebo after 4-weeks washout period.
  Interventions: Drug: ATP mixed probiotics
- Group B (Placebo Comparator): Group B received placebo medication for 6 weeks followed by a crossover to 6 weeks of active medication (ATP mixed probiotics) after 4-weeks washout period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATP mixed probiotics — - Patients in Group A will receive ATP mixed probiotics for 6 weeks. And after 4 weeks wash-out period, they will receive placebo for 6 weeks
  Other Names: DUOLAC
  Arms: Group A
Drug: Placebo — - Patients in Group B will receive placebo for 6 weeks. And after 4 weeks wash-out period, they will receive ATP mixed probiotics for 6 weeks
  Other Names: DUOLAC
  Arms: Group B

SUMMARY:
There is not enough evidence to support the use of probiotics for prevention or treatment of AD in children in clinical practice.

The purpose of this study is to determine whether probiotics is effective in the treatment of atopic dermatitis with cow milk allergy.

ELIGIBILITY:
Inclusion Criteria:

* Under the 2 years old, 36 children
* Mild to moderate atopic dermatitis with cow milk allergy
* Volunteers who agreed by their parents.
* The severity of their disease was assessed by modified SCORAD index

Exclusion Criteria:

* Severe atopic dermatitis
* Patients on systemic steroids, immune-suppression or Korean herbal medicine during the previous 6 weeks
* Anaphylaxis, Angioedema, or severe allergic reaction to the cow milk
* Chronic diarrhea

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Check SCORAD index for severity of atopic dermatitis, symptom diary, blood cytokine and chemokine (IL-4,IL-6, IL-10, IL-13, total IgE, IFN-γ, TGF-β, TNF-α, and IgG4) after drug administration | 6 weeks after patient recruitment

SECONDARY OUTCOMES:
Check SCORAD index for severity of atopic dermatitis, symptom diary, blood cytokine and chemokine (IL-4,IL-6, IL-10, IL-13, total IgE, IFN-γ, TGF-β, TNF-α, and IgG4) after drug administration | 6 weeks after wash-out period

CONTACTS AND LOCATIONS:
Overall Officials: Bok Yang Pyun, Study Chair — Pediatric Allergy & Respiratory Center, Department of Pediatrics, Soonchunhyang University Hospital